CLINICAL TRIAL: NCT05214170
Title: Physician Acceptance of the NeuTrace System for Cardiac Electroanatomic Mapping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuTrace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NT001
Record Dates: First submitted 2021-12-13; First posted 2022-01-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter
Keywords: Cardiac Arrhythmias; Atrial Fibrillation; Atrial Flutter; Electroanatomic Mapping
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, single-arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Electroanatomic mapping with NeuTrace System (Experimental): Patients with arrhythmias undergo electroanatomic mapping with the NeuTrace System.
  Interventions: Device: Electroanatomic mapping with the NeuTrace System

INTERVENTIONS:
Device: Electroanatomic mapping with the NeuTrace System — Patients with arrhythmias undergo electroanatomic mapping with the NeuTrace System.

SUMMARY:
The trial is a prospective, non-randomized, single-arm feasibility trial to evaluate physician acceptance of the NeuTrace System v1.0 for cardiac electroanatomic mapping.

DETAILED DESCRIPTION:
Arrhythmias, or abnormal heart rhythms, are a major cause of morbidity and mortality worldwide. In patients with arrhythmias, electrophysiology (EP) studies are often performed to assess the electrical system of the heart. Since its introduction in the 1990s, electroanatomic mapping has become a cornerstone of EP studies. Electroanatomic mapping systems allow for non-fluoroscopic navigation of the heart and the creation of three-dimensional (3D) anatomic and electroanatomic maps. These maps facilitate diagnosing and treating arrhythmias.

The NeuTrace System is a cardiac EP mapping system that is intended to be used during catheter-based atrial and ventricular mapping procedures. The system is designed to acquire and analyze data points and use this information to display 3D anatomical and electroanatomic mapping of the human heart. The system is used with a compatible, marketed magnetic sensor-enabled catheter and compatible EP recording system to acquire the location information and local electrogram needed to create the cardiac maps. The purpose of the trial is to evaluate physician acceptance and feasibility of the NeuTrace System v1.0 for cardiac electroanatomic mapping.

ELIGIBILITY:
Inclusion Criteria:

* Patient with standard indications for an electrophysiology study and/or catheter ablation per European Heart Rhythm Association/Heart Rhythm Society) guidelines and/or judgement of the investigator
* Age 18 to 80
* Signed Informed Consent Form

Exclusion Criteria:

* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention/percutaneous transluminal coronary angioplasty, or coronary artery stenting which occurred during the 90-day interval preceding the date that participant signed the Informed Consent Form
* Unstable angina
* NHYA class III or IV congestive heart failure and/or known left ventricular ejection fraction less than 45%
* Thrombocytosis, thrombocytopenia
* Contraindication to anticoagulation therapy
* Active systemic infection
* Cryoglobulinemia
* Known reversible causes of arrhythmia
* Any cerebral ischemic event (stroke or transient ischemic attacks) which occurred during the 180-day interval preceding the date the participant signed the Informed Consent Form, or any known unresolved complications from the previous stroke/transient ischemic attack
* Pregnancy
* Unwilling or unable to comply fully with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-05-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Physician rating of the electroanatomic map created by the NeuTrace System via a questionnaire | Immediately post-procedure
  At the completion of each electrophysiology study, the principal investigator will be asked to complete a questionnaire in which he or she qualitatively rates the electroanatomic map created by the NeuTrace System on a numeric scale from 1 to 5 (1 = not satisfied, 5 = very satisfied).

SECONDARY OUTCOMES:
Physician rating of catheter visibility during electroanatomic mapping with NeuTrace System via a questionnaire | Immediately post-procedure
  At the completion of each electrophysiology study, the principal investigator will be asked to complete a questionnaire in which he or she qualitatively rates the visibility of the catheter during electroanatomic mapping with the NeuTrace System on a numeric scale from 1 to 5 (1 = not satisfied, 5 = very satisfied).
Physician rating of the accuracy of the anatomical map created with the NeuTrace System compared to an image obtained via computerized tomography, magnetic resonance imaging, or intracardiac echocardiography via a questionnaire | Immediately post-procedure
  Each participant will have an image obtained of their heart either pre-procedurally via computed tomography or magnetic resonance imaging, or intraprocedurally via intracardiac echocardiography. At the completion of each electrophysiology study, the principal investigator will be asked to complete a questionnaire in which he or she qualitatively rates the accuracy of the electroanatomic map created by the NeuTrace System with the image of the heart obtained via computerized tomography, magnetic resonance imaging, or intracardiac echocardiography.
Measurement of the shift in the electroanatomic during the procedure with the NeuTrace System | Immediately post-procedure
  Shift refers to the movement of an electroanatomic map during the procedure (e.g., the patient moves in relation to the magnetic field). During each electrophysiology study, the principal investigator will annotate a point on the electroanatomic map with the NeuTrace System (X at time 1). The principal investigator will return to and again annotate that same point on the electroanatomic map 20 minutes later (X at time 2). The location of the point will be confirmed via intracardiac echocardiography. The distance between the points (X at time 1 and X at time 2) will be measured on the NeuTrace System in millimeters.
Measurement of the drift in the electroanatomic during the procedure with the NeuTrace System | Immediately post-procedure
  Drift refers to the movement of an electroanatomic map during the procedure due to interference with the magnetic field. During each electrophysiology study, the principal investigator will annotate a point on the electroanatomic map with the NeuTrace System (X1). The principal investigator will then move the X-ray image intensifier (a common source of interference) to a fixed interval above the magnetic field generator and again annotate that same point on the electroanatomic map (X2). The distance between the points (X1 and X2) will be measured on the NeuTrace System in millimeters.
Physician rating of the manual annotation of ablation points with the NeuTrace System via a questionnaire | Immediately post-procedure
  At the completion of each electrophysiology study, the principal investigator will be asked to complete a questionnaire in which he or she qualitatively rates the manual annotation of ablations points during electroanatomic mapping with the NeuTrace System on a numeric scale from 1 to 5 (1 = not satisfied, 5 = very satisfied).
Physician rating of the total mapping time with the NeuTrace System via a questionnaire | Immediately post-procedure
  Total mapping time refers to the time taken to create an electroanatomic map. At the completion of each electrophysiology study, the principal investigator will be asked to complete a questionnaire in which he or she qualitatively rates the total mapping time with the NeuTrace System on a numeric scale from 1 to 5 (1 = not satisfied, 5 = very satisfied).
Number of participants with serious adverse events at 30-day post-procedure telephone follow up | 30 days post-procedure
  Each participant will have a telephone follow-up at 30 days post-procedure for monitoring of serious adverse events. The number of participants with a serious adverse events will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Gediminas Rackauskas, MD, Principal Investigator — Vilnius University Hospital Santaros Klinikos
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No